CLINICAL TRIAL: NCT06846827
Title: A Randomised Controlled Trial to Investigate the Cognitive, Mood, Anti-inflammatory and Metabolic Effects of Chronic Oyster Mushroom Intervention in Older Adults (OYSCOG)
Brief Title: Cognitive, Mood, Anti-Inflammatory and Metabolic Effects of Chronic Oyster Mushroom Intervention in Older Adults
Acronym: OYSCOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Mushroom Council (Other)
Responsible Party: Principal Investigator, Prof Claire Williams, Professor of Neuroscience, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023-088-CW
Record Dates: First submitted 2025-02-20; First posted 2025-02-26 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Cognitive Change; Mood; Metabolism; Inflammatory Response; Weight Change
Keywords: Episodic memory; Executive function; Working memory; Attention; Motor function; Mood; Metabolism; Inflammation
MeSH Terms: conditions — Body Weight Changes; Inflammation | interventions — pleurotolysin B, oyster mushroom; maltodextrin

STUDY DESIGN:
Intervention Model Description: Between- and within-groups (mixed) model
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oyster mushroom (Experimental): dried oyster mushrooms
  Interventions: Other: Oyster mushroom
- Placebo (Placebo Comparator): maltodextrin
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Other: Oyster mushroom — Sachet containing the equivalent of 1 serving (9.39g) of dried ergothioneine-rich Pleurotus oyster mushrooms
  Arms: Oyster mushroom
Other: Maltodextrin — Sachet containing 6.67g of maltodextrin
  Arms: Placebo

SUMMARY:
The Pleurotus oyster species is a common edible mushroom rich in phytochemicals such as proteins, phenolic compounds, dietary fibre and is also particularly rich in ergothioneine, a bioactive known for its neurocognitive benefits. Current research suggests that a mushroom-rich diet may be associated with a lower incidence of age-related neurological disorders, as well as an improvement in the domains of memory and mood.

This randomized double-blind parallel trial investigates the chronic effect (12-weeks) of the equivalent 1 portion of ergothioneine-rich Pleurotus oyster mushrooms (in freeze-dried powdered form), consumed 4 times per week, on cognition and mood, with examination of the potential inflammatory, metabolic, and neurological related mechanisms that may underlie these effects.

DETAILED DESCRIPTION:
The Pleurotus oyster species is a common edible mushroom rich in ergothioneine, a bioactive compound with known neurocognitive benefits. The aim of the OYSCOG trial is to investigate the chronic effect (12-weeks) of the equivalent 1 portion of ergothioneine-rich Pleurotus oyster mushrooms (in dried powdered form), consumed 4 times per week, on cognition and mood, with examination of the potential inflammatory, metabolic, and neurological related mechanisms that may underlie these effects.

A power calculation based on similar research investigating the chronic benefits of other mushroom interventions on cognitive function suggests that 72 participants should give sufficient statistical power (with a=0.05, beta=0.80, cohen's d=0.60). This calculation was based on the average cohen's d value obtained from 7 RCTs examining the effect of Lion's Mane, Reishi mushroom or vitamin D enriched mushroom on global cognitive performance. To allow for a 10% attrition rate, 80 healthy older adults aged 60-80 years old will be recruited. Given the parallel design of the RCT, the cohort will be half split to receive either the control maltodextrin intervention (N=40) or the oyster mushroom intervention (N=40).

During this 12-week RCT, participants will attend the University of Reading, Psychology department on three separate occasions. Specifically, in the pre-screening phase, to check for eligibility, the participants interested in our study will be sent a link to REDCap containing online versions of a Health and Lifestyle Questionnaire containing basic demographic questions and the Epic Norfolk Food Frequency Questionnaire (FFQ), to assess their habitual dietary intake. Then, participants, will be contacted to attend a 3-hour familiarisation session at our department, during which the participant's weight, height and blood pressure will be checked, along with a finger-prick, to ensure that the participants are not anaemic. Furthermore, participants will complete the Raven's Progressive Matrices (RPM) measure of fluid intelligence and will perform each of the cognitive battery tasks twice to control for practice effects in the run up to the test session days.

One week after the familiarisation visit, each participant will attend for the baseline test visit, where they will be asked to complete the battery of cognitive and mood tasks and to have their blood pressure and body weight measured. A few participants (n=40, n=20 from each treatment arm) will also be invited to wear an EEG cap using the Brain Products EEG system with 16 channel active electrodes in order to record EEG measurements while performing a simple computerised cognitive task (N-back task) and while resting with eyes open and eyes closed. EEG spectral activity and event-related potential (ERP) data relating to P300 and N200 peaks will be analysed. Finally, a blood test will be performed at the end of the visit. Following the blood draw, the serum will be separated via centrifuge and stored at -80°C until analysis is complete. Blood serum will be analysed for anti-inflammatory and metabolic ability by measuring the levels of fasting lipids (e.g. total cholesterol) and the markers of inflammation (eg cytokines, interleukins), as well as the levels of the brain derived neurotrophic factor (BDNF), a signalling protein known to be related to neuronal signalling and memory function.

At the end of the baseline visit, participants will receive a 12-week supply of sachets containing either maltodextrin or oyster mushroom, depending on their treatment group allocation. They will be asked to consume one sachet 4 times per week for 12-weeks, to be combined with their usual meals. On the 84th day (week 12), participants will be asked to attend the laboratory for their post-visit test day where they will complete the same test procedures as during the baseline visit. Also, at the end of the post-visit day, participants will be asked to complete two dietary surveys: the Epic Norfolk Food Frequency Questionnaire (FFQ), and a brief dietary questionnaire consisting of specialised questions relating to their habitual mushroom intake.

All test visits will take place in the morning, starting between 9am and 10am and finishing before lunchtime. Participants will be asked to follow a low flavonoid diet for 24 hours in advance of each testing visit. Also, they will be asked to consume a standardised breakfast of lightly buttered toast before attending each test visit.

In terms of the mood and cognitive tests, there will be two cognitive test sessions taking place at the familiarisation visit, one at the baseline visit, and then one at the 12-week post-intervention visit, to assess participants' episodic and working memory, psychomotor and executive function and mood domains. Different versions of the cognitive battery will be used at each presentation to minimise learning, and all versions will be matched for difficulty. The mood and cognitive tests will be completed on a computer and should take no longer than 50-60 minutes to complete. The battery will contain the following tasks:

* Positive and Negative Affect Schedule (PANAS-X)- In this mood task, participants are asked to rate their emotion on a 5-point Likert scale, in response to negative emotions (e.g., guilt, fear), positive emotions (e.g., attentiveness, joy) and other affective states (e.g., surprise, shyness).
* Depression, Anxiety and Stress Scale - 21 items (DASS-21)- This 21-item measure assesses symptoms of depression, anxiety and stress. Each item is scored from 0-3 where higher scores indicate higher levels of distress in anxiety (scores range from 0 to >20), depression (0 to >28) and/or stress (0 to >34).
* Rey Auditory Verbal Learning Task (RAVLT)- This episodic memory task consists of 5 consecutive free recalls of the same 15 nouns presented as an auditory list (list A), followed by recall of a further 15 nouns presented as an interference list (list B) which is recalled only once. List A is subsequently recalled straight after list B and then again after a longer delay of around 30 minutes.
* Task Switching Task (TST) - In this executive function task, participants view 8 spaced radii of a circle above and below a bold line and a stimulus digit selected from 1-9 (except 5) appears clockwise in each segment, either above or below the bold line. Depending on the stimulus position in the segments, participants perform different tasks with each being switched every 4 trials.
* Corsi block tapping task (CBTT)- In this spatial working memory task, participants are shown 9 arranged blocks positioned on a computer screen and are asked to reproduce a given sequence by clicking on the blocks (using the mouse) in the same sequence as they see them.
* Simple and complex finger tapping task (SFT & CFT)- In this psychomotor function task, participants tap on a key as quickly as possible with the index finger of their dominant hand for 1 minute. They then tap out a specific sequence using 4 fingers, again for 1 minute.
* RAVLT word recognition- In this delayed memory task, participants are shown a sequential list of 50 nouns containing the words from lists A and B from the previously described RAVLT task plus 20 additional words not previously heard, and are asked to indicate those from list A.
* N-back (0-Back & 1-Back versions)- In this working memory and attention task, participants are shown a series of stimuli and they have to respond whether the stimuli match or not the target presented at the beginning of the task. For a subset of participants (n=40), this task will be performed while also taking EEG measurements (using Brain Products software and 16 active electrodes), to examine changes in brain activity in response to the target and non-target trials.
* Subjective mental fatigue- At the end of the cognitive battery participants are asked to rate their mental fatigue level on a 9-point Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 60-80 years old
* Have normal vision and hearing
* Have a Body mass index (BMI<=30)
* Have healthy status

Exclusion Criteria:

* Smokers
* Vegans/vegetarians
* Being diagnosed with a psychiatric/neurological condition (eg., stroke, schizophrenia, depression, cognitive impairement, dementia)
* Being diagnosed with a learning/behavioural disorder (e.g. dyslexia, autism, ADHD)
* Being diagnosed with a metabolic disease (eg., type I/II diabetes and cardiovascular disease), or suffer from unmediated hypertension or thrombosis related disorders, or suffer from cancer, kidney or liver disease
* Being anaemic
* Taking disease medication such as anticoagulants, antiplatelet medication, dementia medication, antidepressants, antiepileptic medication, thyroid medication
* Refusing to stop taking vitamin supplements (including prebiotics/probiotics) during the 12-week testing period
* Have food allergies
* Having a difficulty in completing computer-based cognitive tasks

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Affect Schedule (PANAS-X) performance | Baseline and 12-weeks
  A validated self-report measure of affective state. The PANAS comprises of two distinct affective states (positive and negative), as well as 11 individual affective states (fear, guilt, sadness, surprise, hostility, shyness, joviality, self-assurance, attentiveness, fatigue and serenity). Subjects use a likert scale from 1 - 5 to indicate how the word relates to how they are currently feeling. As this analysis is exploratory all affective states will be explored.
Change in Immediate Word Recall performance from the Rey Auditory Verbal Learning Task (RAVLT) | Baseline and 12-weeks
  This episodic memory task consists of 5 consecutive free recalls of the same 15 nouns presented as an auditory list (list A), followed by recall of a further 15 nouns presented as an interference list (list B) which is recalled only once. List A is subsequently recalled straight after list B and then again after a longer delay of around 30 minutes.
Change in the Task Switching Task (TST) performance | Baseline and 12-weeks
  In this executive function task, participants view 8 spaced radii of a circle above and below a bold line and a stimulus digit selected from 1-9 (except 5) appears clockwise in each segment, either above or below the bold line. Depending on the stimulus position in the segments, participants perform different tasks with each being switched in every 4 trials. A response of higher or lower than 5 is made for trials below the bold line, and even or odd for numbers above the line. Outcome measures include overall accuracy and reaction time (RT) on correct trials, as well as accuracy and RT on trials where there is a 'switch cost' from stimuli moving from below to above the bold line and vice versa.
Change in Corsi Block Tapping Test (CBTT) performance | Baseline and 12-weeks
  In this spatial working memory task, participants are shown with 9 arranged blocks positioned on a computer screen and are asked to reproduce a given sequence by clicking on the blocks (using the mouse) in the same sequence as they see them.
Change in Simple Finger Tapping Task (SFTT) performance | Baseline and 12-weeks
  In this motor function task, participants tap on a key (eg the letter C) as quickly as possible with the index finger of their dominant hand for 1 minute.
Change in Complex Finger Tapping Task (CFTT) performance | Baseline and 12-weeks
  In this motor function task, participants tap a specific sequence using 4 fingers, for 1 minute.
Change in RAVLT - Delayed Word Recall performance | Baseline and 12-weeks
  After a period of time participants are asked to recall as many words as possible from list A.
Change in RAVLT - Word Recognition performance | Baseline and 12-weeks
  Following the delayed word recall, words from list A, list B and novel words are displayed sequentially on the screen and participants are asked to indicate which words were from list A only.
Change in Mental Fatigue | Baseline and 12-weeks
  Participants are asked to rate in a 9-point Likert scale their mental fatigue levels, ranging from 1: "Not at all mentally fatigued" to 9: "Extremely mentally fatigued".
Change in 0-Back & 1-Back tasks | Baseline and 12-weeks
  The 0-Back & 1-Back tasks are part of the N-back task that is a measure of working memory where participants are instructed to monitor a series of stimuli and to respond whenever a stimulus is presented that is the same as the one presented n trials previously. Data will be analysed for both accuracy and reaction time on correct trials. For a subset of participants, this task will be conducted while recording EEG in order to monitor change in brain activity in response to target trials.

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure | Baseline and 12-weeks
  Average (triplicate) resting brachial left arm cuffed systolic blood pressure mmHg.
Change in Diastolic Blood Pressure | Baseline and 12-weeks
  Average (triplicate) resting brachial (left arm) cuffed diastolic blood pressure mmHg.
Change in Heart Rate | Baseline and 12-weeks
  Average (triplicate) resting brachial (left arm) cuffed heart rate (beats/minute).
Change in Body Mass Index (BMI) | Baseline and 12-weeks
  Average (triplicate) body mass index (BMI).
Change in neurotrophic marker | Baseline and 12-weeks
  Blood serum levels of the Brain Derived Neurotrophic Factor (BDNF).
Change in metabolic markers | Baseline and 12-weeks
  Blood serum levels of glucose & triglycerides (TAG).
Change in inflammatory markers | Baseline and 12-weeks
  Blood serum levels of nitrite, nitric oxide (NOX), inducible nitrous oxide synthase (iNOS), cyclooxygenase-2 (COX-2) and Interleukin-6 (IL-6).
Change in P300 | Baseline and 12-weeks
  The ERP measure of P300 latency and amplitude will be assessed using EEG (electroencephalography) in a subset of participants during resting state (eyes open and closed) and during the 0-Back & 1-Back tasks.
Change in N200 | Baseline and 12-weeks
  The ERP measure of N200 latency and amplitude will be assessed using EEG (electroencephalography) in a subset of participants during resting state (eyes open and closed) and during the 0-Back & 1-Back tasks.
Change in Power Spectral Density (PSD) | Baseline and 12-weeks
  The PSD for Alpha, Beta, Gamma, Delta, and Theta bands will be examined during at the resting state (eyes open/eyes close) and while performing the N-Back task.

OTHER OUTCOMES:
Health and Lifestyle Questionnaire | Baseline
  The online Health and Lifestyle questionnaire includes basic demographic questions to screen participants.
Epic-Norfolk Food Frequency Questionnaire (FFQ) | Baseline
  Epic-Norfolk Food Frequency Questionnaire is an online validated tool to assess participants' habitual dietary intake of different foods including fruits, vegetables, pasta, bread, meat, fish, dairy, sweets, sauces and drinks. Participants will be required to stipulate their intake frequency of individual foods from nine options from never to more than 6 portions/day. The FETA analytical tool will be used to estimate the daily fruit and vegetable intake.
Epic-Norfolk Food Frequency Questionnaire (FFQ) | 12-weeks
  Epic-Norfolk Food Frequency Questionnaire is an online validated tool to assess participants' habitual dietary intake of different foods including fruits, vegetables, pasta, bread, meat, fish, dairy, sweets, sauces and drinks. Participants will be required to stipulate their intake frequency of individual foods from nine options from never to more than 6 portions/day. The FETA analytical tool will be used to estimate the daily fruit and vegetable intake.
Specialised dietary survey | 12-weeks
  Short survey relating to mushroom habitual intake.

CONTACTS AND LOCATIONS:
Overall Officials: Claire M Williams, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All personally related collected information will be kept in locked filing cabinets in the Nutritional Unit of the School of Psychology. The digital health questionnaires used for the purpose of pre-screening participants as well as any digital research data will be stored in the Research Electronic Data Capture (REDCap) database, stored on the University secure network cloud.
  All relevant study outcomes described in the Ethics Review Application Form (including the demographic and anthropometric data (such as age, sex, BMI, blood pressure) as well as the performance scores of the battery tests assessing cognitive function and mood and the results of the blood tests measuring immunological and metabolic function) will be preserved and made available in anonymised form.

REFERENCES:
- [Background] Li IC, Chang HH, Lin CH, Chen WP, Lu TH, Lee LY, Chen YW, Chen YP, Chen CC, Lin DP. Prevention of Early Alzheimer's Disease by Erinacine A-Enriched Hericium erinaceus Mycelia Pilot Double-Blind Placebo-Controlled Study. Front Aging Neurosci. 2020 Jun 3;12:155. doi: 10.3389/fnagi.2020.00155. eCollection 2020. PMID 32581767
- [Background] Mori K, Inatomi S, Ouchi K, Azumi Y, Tuchida T. Improving effects of the mushroom Yamabushitake (Hericium erinaceus) on mild cognitive impairment: a double-blind placebo-controlled clinical trial. Phytother Res. 2009 Mar;23(3):367-72. doi: 10.1002/ptr.2634. PMID 18844328
- [Background] Saitsu Y, Nishide A, Kikushima K, Shimizu K, Ohnuki K. Improvement of cognitive functions by oral intake of Hericium erinaceus. Biomed Res. 2019;40(4):125-131. doi: 10.2220/biomedres.40.125. PMID 31413233
- [Background] Tsuk S, Lev YH, Rotstein A, Carasso R, Zeev A, Netz Y, Dwolatski T, Steiner G. Clinical Effects of a Commercial Supplement of Ophiocordyceps sinensis and Ganoderma lucidum on Cognitive Function of Healthy Young Volunteers. Int J Med Mushrooms. 2017;19(8):667-673. doi: 10.1615/IntJMedMushrooms.2017021202. PMID 29199566
- [Background] Wang GH, Wang LH, Wang C, Qin LH. Spore powder of Ganoderma lucidum for the treatment of Alzheimer disease: A pilot study. Medicine (Baltimore). 2018 May;97(19):e0636. doi: 10.1097/MD.0000000000010636. PMID 29742702
- [Background] Zajac IT, Barnes M, Cavuoto P, Wittert G, Noakes M. The Effects of Vitamin D-Enriched Mushrooms and Vitamin D3 on Cognitive Performance and Mood in Healthy Elderly Adults: A Randomised, Double-Blinded, Placebo-Controlled Trial. Nutrients. 2020 Dec 16;12(12):3847. doi: 10.3390/nu12123847. PMID 33339304
- [Background] Grozier CD, Alves VA, Killen LG, Simpson JD, O'Neal EK, Waldman HS. Four Weeks of Hericium erinaceus Supplementation Does Not Impact Markers of Metabolic Flexibility or Cognition. Int J Exerc Sci. 2022 Oct 1;15(2):1366-1380. doi: 10.70252/XZKO8571. eCollection 2022. PMID 36582308

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT06846827/Prot_SAP_000.pdf